CLINICAL TRIAL: NCT06312787
Title: A Phase 1, Open-label, Randomized, Crossover Study to Evaluate the Relative Bioavailability and Food Effect of a Tablet Formulation of VX-118 in Healthy Adult Subjects
Brief Title: A Study to Evaluate the Relative Bioavailability and Food Effect of a VX-118 Tablet Formulation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: VX23-118-002
Record Dates: First submitted 2024-03-08; First posted 2024-03-15 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Sequence 1 (Experimental): Participants will receive a single dose of VX-118 as a suspension in the fasted state in dosing period 1, followed by a single dose of VX-118 as tablets in the fasted state in dosing period 2, followed by a single dose of VX-118 as tablets in the fed state in dosing period 3. A washout period of 8 days will be maintained between the 3 dosing periods.
  Interventions: Drug: VX-118
- Sequence 2 (Experimental): Participants will receive a single dose of VX-118 as tablets in the fasted state in dosing period 1, followed by a single dose of VX-118 as tablets in the fed state in dosing period 2, followed by a single dose of VX-118 as a suspension in the fasted state in dosing period 3. A washout period of 8 days will be maintained between the 3 dosing periods.
  Interventions: Drug: VX-118
- Sequence 3 (Experimental): Participants will receive a single dose of VX-118 as tablets in the fed state in dosing period 1, followed by a single dose of VX-118 as a suspension in the fasted state in dosing period 2, followed by a single dose of VX-118 as tablets in the fasted state in dosing period 3. A washout period of 8 days will be maintained between the 3 dosing periods.
  Interventions: Drug: VX-118

INTERVENTIONS:
Drug: VX-118 — Tablets and Suspension for Oral Administration

SUMMARY:
The purpose of this study is to evaluate the relative bioavailability, effect of food on the pharmacokinetic parameters, and safety and tolerability, of a tablet formulation of VX-118 in healthy participants.

DETAILED DESCRIPTION:
This clinical trial information was submitted voluntarily under the applicable law and, therefore, certain submission deadlines may not apply. (That is, clinical trial information for this applicable clinical trial was submitted under section 402(j)(4)(A) of the Public Health Service Act and 42 CFR 11.60 and is not subject to the deadlines established by sections 402(j)(2) and (3) of the Public Health Service Act or 42 CFR 11.24 and 11.44.).

ELIGIBILITY:
Key Inclusion Criteria:

* Body mass index (BMI) of 18.0 to 32.0 kilogram per meter square (Kg/m^2), both inclusive
* A total body weight greater than (>) 50 kg
* Participants of non-childbearing potential

Key Exclusion Criteria:

* History of febrile illness or other acute illness that has not fully resolved within 14 days before the first dose of study drug
* Any condition possibly affecting drug absorption
* Hypersensitivity to any component of the investigational drug product

Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2024-04-02 (Actual); Primary Completion 2024-05-04 (Actual); Study Completion 2024-05-04 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of VX-118 | Pre-dose up to 192 hours Post-dose
Area Under the Concentration Versus Time Curve (AUC) of VX-118 | Pre-dose up to 192 hours Post-dose

SECONDARY OUTCOMES:
Safety and Tolerability as Assessed by Number of Participants With Adverse Events (AEs) | Day 1 up to Day 27

CONTACTS AND LOCATIONS:
Locations (1):
- Celerion - Lincoln, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent-research/clinical-trial-data-sharing